CLINICAL TRIAL: NCT05546203
Title: The Effectiveness of Trigger Point Treatment in Chronic Pelvic Pain; A Pilot Randomized Controlled Trail
Brief Title: Trigger Point Treatment in Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Munzur University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Kubra Sagır, Research Assistant, Munzur University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kubra_2018
Record Dates: First submitted 2022-09-16; First posted 2022-09-19 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Chronic Pelvic Pain Syndrome; Myofascial Trigger Point Pain
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Acupressure; Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Randomized parallel designed two arm clinical study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ischemic compression (IC) group (Experimental): Ischemic compression group received ischemic compression and standardized exercise program twice a week for 6 weeks. Each session takes 50 minutes.
  Interventions: Other: Ischemic compression; Behavioral: Standardized exercise program
- Low-level laser therapy (LLLT) group (Experimental): Low-level laser therapy group received Low-level laser therapy and standardized exercise program twice a week for 6 weeks. Each session takes 50 minutes.
  Interventions: Device: Low-level laser therapy; Behavioral: Standardized exercise program

INTERVENTIONS:
Other: Ischemic compression — IC was applied over the detected MTrPs and the participant was asked to describe the pressure and pain she felt . It was started with moderate tolerable pressure (7/10) and then severity was increased. The color of the thumb pulp was observed to control the pressure. The pressure was continued for 90 sec. The patient's pain sensation continued to be questioned and the pressure was controlled to a level at "comfortable pain"
  Arms: Ischemic compression (IC) group
Device: Low-level laser therapy — LLLT was applied for 90 sec at each MTrPs with a frequency of 2000 Hz (3 J) using a GaAs diode laser instrument (Roland Serie Elettronica Pagani, wavelength 904 nm, the frequency range of 5-7000 Hz and maximum peak power of 27, 50 or 2764 W) . The laser probe was held perpendicular to the MTrPs in skin contact without pressure.
  Arms: Low-level laser therapy (LLLT) group
Behavioral: Standardized exercise program — The standardized exercise program included stretching and pilates exercises for core stabilization. All exercises were supervised by the same physiotherapist whom certificated by The Australian Physiotherapy and Pilates Institute (APPI). Pilates exercises were selected from APPI's mat-work exercises and performed in accordance with APPI principles. In addition, patients performed stretching exercises for 5 days a week and pilates exercises for 3 days a week at home.

SUMMARY:
Objective: To investigate the effectiveness of ischemic compression and low-level laser therapy methods combined with exercise on the myofascial trigger points in women with Chronic Pelvic Pain and to determine which method is more effective.

Methods: It was a parallel designed, single-blind pilot randomized clinical trial. Patients were enrolled in the Department of Obstetrics and Gynecology (at Istanbul University-Cerrahpasa). The patients were diagnosed by a gynecologist (F.G.U and C. Y.), referred to the clinical laboratory of physiotherapy and rehabilitation to participate (by physiotherapists K.S. and E.K.M.) in the trial from September 2017 to June 2019. Twenty-eight women patients with Chronic Pelvic Pain were included into the trial. Patients were randomized into two groups. Group 1 received ischemic compression and Group 2 received low-level laser therapy twice a week for 6 weeks. Both groups received the same standard exercise program. Pain, range of motion, pelvic floor symptom severity, quality of life, satisfaction, anxiety, and depression were assessed after 6 weeks and 1-year follow up.

DETAILED DESCRIPTION:
Chronic pelvic pain (CPP) is chronic or persistent pain perceived in structures related to the pelvic region. CPP prevalence range between 5.7 % and 26.6 % in women. CPP is associated with symptoms suggestive of the lower urinary tract, sexual, bowel, pelvic floor, or gynecological dysfunction. It is often associated with negative emotional consequences and impaired quality of life (QoL) Analgesics, hormone therapy, physiotherapy, psychological treatment, and surgical methods are widely used in the treatment of CPP. Medications provide pain and visceral management, surgery provides correction of structure, but physiotherapy approachs provides functional restoration. Musculoskeletal pelvic pain is commonly originated myofascial, musculoskeletal, neuromuscular structures. CPP patients have myofascial trigger points (MTrPs) located in the lower back, abdominal wall, and pelvic girdle, which may be the primary source of pain. These MTrPs are usually located in levator ani, obturator internus, piriformis, gluteal muscles, quadratus lumborum and abdominal wall muscles. The MTrPs are hyperirritable spots within a taut band, activated by repeated or chronic muscular overload.

Ischemic compression (IC), in the other words trigger point compression, is an effective method in the treatment of MTrPs in many musculoskeletal problems. IC changes the circulatory perfusion of skin and is especially valuable in muscles that are not suitable for stretch. It is less common to use pelvic floor rehabilitation, urological CPP, interstitial cystitis and painful bladder syndrome and CPP yet. Low-level laser therapy (LLLT) reduces pain in MTrPs lead to musculoskeletal system disorders. LLLT increases oxygen supply to hypoxic cells in MTrPs areas by regulating microcirculation as well as it has analgesic, biostimulation, and wound healing effects . In the literature, it is seen that IC and LLLT are effective on MTrPs, and IC is used in pelvic pain in a few studies. But the use of LLLT in pelvic pain has not been found. It is a known fact that exercise is the basis for these MTrPs treatments. In light of this knowledge, investigetors hypothesized that both IC and LLLT combined with exercise would be an effective methods in the management of CPP.

ELIGIBILITY:
Inclusion Criteria:To be eligible,

* participants had to be between 18-50 years of age,
* had pain/discomfort in the lower abdominal and pelvic region lasting for 3 months in the last 6 months.
* Patients with MTrPs in at least two of the examined muscles (rectus abdominis, piriformis, quadratus lumborum, gluteus maximus-medius, adductor magnus, hamstring) were included in order to perform statistical analysis.

Exclusion Criteria: The exclusion criteria were;

* anticoagulation or bleeding disorders,
* neuropathy, central nervous system disorders,
* advanced psychiatric disorders,
* significant pelvic pathology or abnormality, severe prolapse, pregnancy,
* to have undergone major surgery and pelvic surgery with general anesthesia in the last 3 months,
* to have received treatment including electrotherapy and manual therapy for the pelvic region in the last 6 months.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 1- a day before the treatment program 2- at the time of discharge (end of the 6 weeks program) 3- at the 1 year follow-up
  Pain intensity was assessed using the VAS, in which the patients were asked to indicate their perceived pain during rest, activity and at night (0-10 numeric pain rating scale, with 0 as no pain and 10 as worst imaginable pain) .
Pressure Pain Threshold (PPT) | 1- a day before the treatment program 2- at the time of discharge (end of the 6 weeks program) 3- at the 1 year follow-up
  Handheld pressure algometer (Commander Algometer, J Tech Medical Industries, Midvale, Utah; maximum output=111.6N/cm2) was used to measure PPT on the MTrPs determined by clinical examination. Investigetors asked the subjects to say "stop" as soon as a discernible sensation of pain was felt. When the subject lying on loose position, a 1-cm2 algometer probe was placed perpendicularly on the MTrPs, and the pressure was increased gradually (1 lb/s). First painful threshold was recorded, mean value of two measurements, with 3 minutes interval, was used for analysis .

SECONDARY OUTCOMES:
Range of Motion (ROM) | 1- a day before the treatment program 2- at the time of discharge (end of the 6 weeks program) 3- at the 1 year follow-up
  Lumbar spine active ROM from full extension to full flexion, and hip active ROM on flexion, extension and mediolateral rotation was measured using a digital goniometer (Baseline Evaluation Instrument®, Fabrication Enterprises, Inc.). Average of 3 repetitions was recorded for analysis.
The Pelvic Floor Bother Questionnaire (PFBQ) | 1- a day before the treatment program 2- at the time of discharge (end of the 6 weeks program) 3- at the 1 year follow-up
  The Pelvic Floor Bother Questionnaire (PFBQ) was used to identify the presence and degree of bother related to common pelvic floor problems. It had excellent test-retest reliability (0.998, p<0.0001).
Urogenital Distress Inventory (UDI-6) | 1- a day before the treatment program 2- at the time of discharge (end of the 6 weeks program) 3- at the 1 year follow-up
  Urogenital Distress Inventory (UDI-6) was used to assess urinary symptoms related QoL. It consists of 6 questions covering three domains: stress urinary incontinence, detrusor overactivity, bladder outlet obstruction. It had high internal consistency (Cronbach's alpha: 0.74) and test-retest reliability (Spearman's rho:0.99, p<0.001).
Short Form Health Survey-36 (SF-36) | 1- a day before the treatment program 2- at the time of discharge (end of the 6 weeks program) 3- at the 1 year follow-up
  Short Form Health Survey-36 (SF-36) was used to assess the general QoL. It consists of 36 items, 8 sub-scales; physical and social functioning, role limitations due to physical health and emotional problems, emotional well-being, pain, energy-fatigue, general health status. It has recently been shown to be highly reliable (Cronbach alpha value of the subscales varied in the range 0.792-0.992) in chronic pain.
The Hospital Anxiety and Depression Scale (HADS) | 1- a day before the treatment program 2- at the time of discharge (end of the 6 weeks program) 3- at the 1 year follow-up
  The Hospital Anxiety and Depression Scale (HADS) was used to identify the anxiety disorders and depression among patients. It has anxiety and depression subscale, both containing seven items. It had high internal consistency (Cronbach's alpha coefficient: 0.8525 for anxiety subscale and 0.7784 for depression subscale)
Patient Global Impression of Improvement (PGII) | 1- a day before the treatment program 2- at the time of discharge (end of the 6 weeks program) 3- at the 1 year follow-up
  Patient Global Impression of Improvement (PGII) used to assess patient satisfaction. It consists of 7-point question (1=very much better, 7=very much worse) asking the patient's level of recovery after treatment. PGII have a significant correlation with incontinence episode frequency, stress pad test, and incontinence-related quality of life .

CONTACTS AND LOCATIONS:
Overall Officials: Kübra Sağır Ataş, MSC, Principal Investigator — Munzur University
Locations (1):
- Munzur University, Tunceli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Laser therapy and needling in myofascial trigger point deactivation — https://www.jstage.jst.go.jp/article/josnusd/55/2/55_175/_article/-char/ja/
- See also: Anaesthetic injection versus ischemic compression for the pain relief of abdominal wall trigger points in women with chronic pelvic pain. — http://dx.doi.org/10.1186/s12871-015-0155-0